CLINICAL TRIAL: NCT04287673
Title: Associated Disorders of Locomotion and Postural Control of Axial Segments in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRR-2015-1
Record Dates: First submitted 2020-02-05; First posted 2020-02-27 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Trunk control; Postural Control; Cerebral Palsy; Rehabilitation; Axial segments
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RIST-UR (Experimental): Group having performed the rehabilitation involving strongly the trunk for the first 3 months and then having performed its usual rehabilitation for the last 3 months.
  Before and after each 3-months period, an evaluation of the postural control of the trunk (using the Trunk Control Measurement Scale and a dynamic posturography on an unstable sitting device) and a clinical gait analysis were performed.
  Interventions: Other: Rehabilitation involving strongly the trunk
- UR-RIST (Experimental): Group having performed its usual rehabilitation for the first 3 months and then having performed the rehabilitation involving strongly the trunk for the last 3 months.
  Before and after each 3-months period, an evaluation of the postural control of the trunk (using the Trunk Control Measurement Scale and a dynamic posturography on an unstable sitting device) and a clinical gait analysis were performed.
  Interventions: Other: Rehabilitation involving strongly the trunk
- Typically Developing children (No Intervention): Typically developing children who served as a control group in the first assessment (Trunk Control Measurement Scale, dynamic posturography on an unstable sitting device, clinical gait analysis)

INTERVENTIONS:
Other: Rehabilitation involving strongly the trunk — The Rehabilitation involving strongly the trunk (RIST) leaded by a physiotherapist was based on exercises in different postures performed by the child each day that strongly involve the trunk to cope with balance.
  Arms: RIST-UR; UR-RIST

SUMMARY:
Gait abnormalities, which occur in Cerebral Palsy (CP), are characterized usually by a toe-to-floor or a plantar-to-floor initial contact (equinus gait), followed by an early braking of the tibia's forward progression (during ankle dorsiflexion). This causes consequently a trunk deceleration. Moreover, children with CP have difficulties to stabilize the trunk and the head in the space, and that could have impact on gait. If equinus gait is often attributed to the triceps surae spasticity, recent works suggest rather that this early braking of the dorsiflexion could be a motor adaptation to axial postural control difficulties. This thesis project aims firstly to attest that locomotor disorders are related to these difficulties in the stabilization of the axial body segments in children with CP and, secondly, to show that improving the trunk and head postural control with a specific rehabilitation protocol could reduce the early braking of the dorsiflexion and, consequently, the gait abnormalities observed in CP.

ELIGIBILITY:
Inclusion Criteria:

* Gross Motor Function Classification System I or II
* no or minimal contracture of the triceps surae
* presence of soleus spasticity

Exclusion Criteria:

* botulinum toxin injections or surgery in the lower limb respectively in the 6 and 12 months preceding the study
* any modification of the physical or orthopaedic therapy within the last two months
* minimal hip flexion above 20° in a clinical examination
* pain in the lower legs when standing or walking

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change of the peak of ankle negative power during the weight acceptance phase of gait | Change from baseline to the end of the first 3-months period of rehabilitation and from this latter to the end of the second 3-months period of rehabilitation
  In watts per kg.
Change of the peak of trunk's anterior deceleration during the weight acceptance phase of gait | Change from baseline to the end of the first 3-months period of rehabilitation and from this latter to the end of the second 3-months period of rehabilitation
  In m/s²
Change of the peak of the center of mass downward deceleration during the weight acceptance phase of gait | Change from baseline to the end of the first 3-months period of rehabilitation and from this latter to the end of the second 3-months period of rehabilitation
  In m/s²
Change of the score of the Trunk Control Measurement Scale (TCMS) | Change from baseline to the end of the first 3-months period of rehabilitation and from this latter to the end of the second 3-months period of rehabilitation
  Score from 0 to 58. The higher the score, the better the trunk control.
Change of the center of pressure velicoty during unstable sitting posturography | Change from baseline to the end of the first 3-months period of rehabilitation and from this latter to the end of the second 3-months period of rehabilitation
  In mm²/s
Change of the center of pressure sway area during unstable sitting posturography | Change from baseline to the end of the first 3-months period of rehabilitation and from this latter to the end of the second 3-months period of rehabilitation
  In mm²

SECONDARY OUTCOMES:
Change of the Dimensionless walking speed | Change from baseline to the end of the first 3-months period of rehabilitation and from this latter to the end of the second 3-months period of rehabilitation
  Walking speed normalized to the length of the lower limb
Change of the dimensionless step width | Change from baseline to the end of the first 3-months period of rehabilitation and from this latter to the end of the second 3-months period of rehabilitation
  Step width during walking normalized to the width of the pelvis
Change of the center of pressure velicoty during quiet standing | Change from baseline to the end of the first 3-months period of rehabilitation and from this latter to the end of the second 3-months period of rehabilitation
  In mm²/s
Change of the center of pressure sway area during quiet standing | Change from baseline to the end of the first 3-months period of rehabilitation and from this latter to the end of the second 3-months period of rehabilitation
  In mm²

CONTACTS AND LOCATIONS:
Overall Officials: Christian Beyaert, PU-PH, Principal Investigator — University of Lorraine
Locations (1):
- Institut Régional de Médecine Physique et de Réadaptation, Nancy, France